CLINICAL TRIAL: NCT04958512
Title: Clinical Study of Yangxue Qingnao Pill in the Treatment of Mild Vascular Cognitive Impairment Without Dementia (VCIND)
Brief Title: Treatment of Mild Vascular Cognitive Impairment With Yangxue Qingnao Pill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2017154
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Cerebrovascular Diseases
Keywords: cognitive disorder
MeSH Terms: conditions — Cerebrovascular Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- blank control group (Other)
  Interventions: Other: blank control group
- treatment group(Yangxue Qingnao pill) (Experimental)
  Interventions: Drug: Yangxue Qingnao pill
- control group(hidezhen) (Active Comparator)
  Interventions: Drug: Hydergotoxine mesylate tablets

INTERVENTIONS:
Drug: Yangxue Qingnao pill — The treatment group (20 cases) was treated with Yangxue Qingnao pill (2.5g / time, 3 times / day, orally for 6 months
  Arms: treatment group(Yangxue Qingnao pill)
Drug: Hydergotoxine mesylate tablets — The control group (n = 20) was treated with hidezhen 3 mg per day before meals for 6 months
  Arms: control group(hidezhen)
Other: blank control group — There were 20 cases in the blank control group.Outpatient consultation at any time was prescribed.
  Arms: blank control group

SUMMARY:
In this study, the effectiveness of vascular cognitive impairment was compared among the three groups, namely, the xidezhen group, the Yangxue Qingnao pill group and the placebo group

DETAILED DESCRIPTION:
The risk factors of various cerebrovascular diseases (atherosclerosis, stroke, hypertension, coronary heart disease, atrial fibrillation, dyslipidemia, diabetes mellitus) are both risk factors of Alzheimer's disease and one of the many causes of vascular dementia. There are many manifestations of mental retardation caused by cerebrovascular diseases. The most prominent aspect is cognitive and behavioral impairment, which is characterized by mental retardation, forgetfulness, misunderstanding and poor calculation ability. Yangxue Qingnao pill (z20063808:) is produced by Tianshili Pharmaceutical Group Co., Ltd, And then improve the ability of learning and memory. Some clinical application results show that the drug can significantly improve the cognitive and behavioral ability of patients with ischemic stroke, improve the cognitive function of patients with mild Alzheimer's disease, and improve the quality of life. Therefore, this study mainly compared the effectiveness of treatment of vascular cognitive impairment in three groups, namely, the xidezhen group, the yangxueqingnaowan group and the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Over 50 years old, under 85 years old, male and female, including 50 and 85 years old;
2. The patients agreed to participate in the trial and signed the informed consent.
3. The diagnostic criteria for vascular cognitive impairment without dementia are as follows:

   1. There are risk factors of cerebrovascular disease or the existence of cerebrovascular disease;
   2. The development of cognitive impairment was fluctuating;
   3. Mild memory impairment or retention;
   4. There is a causal relationship between cerebrovascular disease and cognitive impairment, and other diseases are excluded;
   5. The activities of daily living remained normal;
   6. According to the diagnostic criteria of mild cognitive impairment (MCI) developed by Xiao Shifu, the subjects' MMSE score was less than or equal to 26

Exclusion Criteria:

1. The researchers considered that it was not suitable to be included in the study;
2. Known liver diseases of clinical significance, which may hinder patients from completing the test, and / or total bilirubin, aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase are 1.5 times higher than the upper limit of normal value;
3. The patients with known clinically significant kidney disease may be prevented from completing the test, and / or the serum creatinine is higher than the normal range in the laboratory, and / or the blood urea nitrogen is 1.5 times higher than the normal range;
4. He had a history of acute cerebrovascular disease within 3 months;
5. At present, there is active epilepsy;
6. History of mental illness;
7. Peptic ulcer and gastrointestinal bleeding;
8. Any of the tested drugs was taken within 28 days before medication, which may cause cognitive changes and important organ damage.
9. Accompanied by unstable blood system and immune system diseases, is not in clinical remission.
10. Malignant tumor or intracranial tumor is known;
11. Those who had surgery within three months or had a history of trauma.
12. There are other advanced, serious or unstable diseases, which affect the evaluation of its efficacy and safety;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Scale (MoCA) | at 6th month
  Level of cognition,ranging from 0-30 points, the higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided